CLINICAL TRIAL: NCT07256574
Title: Sun-Kissed Serenity: Morning Rays for a Brighter Mind
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 37231
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Mental Status Change

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Behavioral: Morning sunlight

INTERVENTIONS:
Behavioral: Morning sunlight — Participants are asked to get 15 minutes of morning sunlight every day for 30 days.

SUMMARY:
Sun-Kissed Serenity: Morning Rays for a Brighter Mind is a 30-day dawn rendezvous with nature. Participants are asked to stand outside for 15 minutes each morning, track progress with surveys, and support mental health with natural light.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to meticulously evaluate the impact of daily morning sunlight exposure on mental well-being over a span of 30 days. In an era where society is increasingly fraught with overstimulation and stress, this study seeks to explore a simple, natural intervention that has been both scientifically and anecdotally linked to improved mental health outcomes. Leveraging the NIH Toolbox® Positive Affect Survey and the Personal Feelings Survey, this online study aims to quantify the effects of a 15-minute morning sunlight exposure routine on participants' mood, stress levels, and overall sense of well-being.

The objective behind this innovative approach is to empower individuals to discover the potential mental health benefits of integrating a brief period of sunlight exposure into their daily morning routine. By participating in this trial, individuals are not only taking an active step towards potentially enhancing their own mental wellness but are also contributing valuable data to a broader scientific endeavor aimed at validating a cost-free, accessible method for supporting mental health.

This study will utilize a variety of validated tools to rigorously assess changes in participants' emotional states and personal well-being throughout the trial period. This includes tracking shifts in positive affect, stress levels, and overall mood, to determine whether this straightforward daily practice can yield significant improvements in mental health metrics.

The significance of this study lies in its potential to offer a low-cost, universally accessible intervention for enhancing mental wellness without the need for pharmaceuticals, subscriptions, or the risk of adverse side effects. Despite variables such as weather conditions or individual daily routines, the prospect of establishing a free, evidence-based practice for reducing stress and elevating mood holds considerable promise. Through this remotely conducted trial, the investigators aim to gather conclusive evidence on the efficacy of morning sunlight exposure as a tool for mental health support, thereby contributing to the development of simple, natural strategies for managing stress and improving emotional well-being in today's fast-paced world.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox® Item Bank v3.0 - Positive Affect Survey (Ages 18+) Score | Change from baseline (Day 1-3) in positive affect scores at 4 weeks after the start of the intervention (Day 28-32)
  This survey assesses your level of positive affect in the past 7 days. Please respond to each question or statement by selecting one option that best describes your feelings or experiences.
Personal Feelings Survey | Change from baseline (Day 1-3) in feelings of isolation scores at 4 weeks after the start of the intervention (Day 28-32)
  This survey aims to understand your personal feelings, particularly about being alone or feeling isolated. You are asked to indicate how often you feel a certain way.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/morning-sunlight-and-mental-health/?nocache=1761163160